CLINICAL TRIAL: NCT06284889
Title: Behavioral Activation for the Treatment of Depression in Older Adults: A Randomised Controlled Multicenter Trial in Primary Care (DepActive)
Brief Title: Behavioral Activation for the Treatment of Depression in Older Adults
Acronym: DepActive
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government); Sormland County Council, Sweden (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DepActive
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: Behavioral activation; Older adults; Activity; Primary care
MeSH Terms: conditions — Depression; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomised controlled multi-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Brief Behavioral Activation
  Interventions: Behavioral: Behavioural activation; Other: Treatment as usual (TAU)
- Treatment as usual (TAU) (Placebo Comparator): Treatment as usual regarding depression received at their primary care centre.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Behavioural activation — Session 1: Face-to-face; Psychoeducation about depression; treatment rationale for Behavioral Activation (BA); rationale and instructions for activity log;
  Session 2: Via telephone; Discussion of life goals and values; planning of activities aligned with life goals and values for coming week
  Session 3: Via telephone; Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for coming week.
  Session 4: Via telephone; Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for the coming week; instructing the participant to independently continue to plan activities for the coming month.
  Session 5: Via telephone; Troubleshooting any problems carrying out activities; reviewing treatment; stressing the importance of continuing to engage in activities aligned with life goals and values; creating a maintenance plan.
  Arms: Treatment
Other: Treatment as usual (TAU) — Treatment as usual regarding depression received at their primary care centre.

SUMMARY:
Depression affects between 5-15% of adults ≥ 65 years in Sweden. Depression in older adults reduces functional ability and quality of life, and increases the risk for morbidity, loneliness, and suicide. Psychological treatment is recommended as a first-line treatment for depression, which about 3% of older adults with depression in Sweden report receiving. One effective psychological treatment is behavioral activation, which reduces depressive symptoms by increasing enjoyable, meaningful and important activities, for example exercise and social activities. The research group conducted a pilot study of telephone based behavioral activation for isolated older adults with depression during the COVID-19 pandemic. The intervention consisted of four telephone calls, and the results showed a significant decrease in depressive symptoms, with maintained effects for six months.

250 individuals will participate in the study. Half of the participants will be randomised to start the intervention immediately, while the other half of the participants will be randomized to a control group receiving treatment as usual at their respective primary care center. Participants will be asked to fill in questionnaires before, after treatment. Questionnaires will also be sent 3- and 6 months after treatment to follow up on the results. Patients will be asked to wear an accelerometer for 5-7 days to record their activity level at baseline, post-intervention and after 3-months. A smaller group of participants (10-15) will be asked to participate in a more detailed interview about how they experienced the treatment.

DETAILED DESCRIPTION:
In Sweden, depression among the elderly is a major public health concern. Major depression occurred in 5-15 % of the older population in Sweden, and one third of the women and a fifth of the men 65 years and older reported subclinical depressive symptoms. Several mental health experts raise concerns that there will be an increase of psychiatric illness during and after COVID-19, particularly among the elderly.

Depression in older individuals can be treated with antidepressant medication, psychological interventions and physical activity. However, the majority of the older individuals state that they would prefer psychological treatments to medication, which poses a challenge during COVID-19 as such treatments are often delivered face-to-face. Psychological treatments delivered via the Internet are as efficacious as face-to-face, but only 3-4% of the individuals 65 years and above in Sweden use digital applications that replace physical healthcare visits.

The purpose of this randomised controlled multicenter study is to evaluate the effects and outcomes of a telephone-delivered Behavioral Activation-treatment for older adults with depression in primary care within the framework of the research project DepActive. Our study specifically aims to: 1. investigate the effect of a telephone-delivered BA-treatment for older adults with depression in primary care with regards to a. depressive symptoms (primary outcome measure) b. depression diagnosis c. anxiety symptoms d. quality of life e. activity level f. functional ability g. cognitive function h. loneliness i. self-efficacy j. cost effectiveness k. care consumption including pharmacological treatment 2. explore patients' and therapists' experiences of the treatment 3. investigate to which extent the BA-treatment corresponds to person-centered care 4. investigate the mediating role of type of activity and level of physical activity with regards to improvement in depressive symptoms 5. investigate whether the intervention impacts the need for community healthcare services for participants utilizing such services.

The study is a multi-center randomised controlled clinical trial in primary care in the Swedish county councils of Vastmanland, Uppsala and Sormland.

Participants will be recruited from multiple primary care centers in each region. If the participant is enrolled in the study, the study therapist performs the randomisation by using an online randomisation software with a 1:1, random-blocks sequence. The participants are randomised consecutively to two arms: control group or intervention group. The control group will receive treatment as usual (TAU) in primary care, and the intervention group will receive TAU with the addition of a five-session telephone-based BA-intervention over an eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* Participants should fulfill criteria for current major depressive episode or sub-threshold depressive episode.
* Eligible participants should be 65 years or older, should be fluent in spoken and written Swedish to understand the treatment materials, have access to telephone, and be interested in participating in the trial.

Exclusion Criteria:

* Severe depression, elevated suicide risk, current substance use disorder, current or previous manic or hypomanic episodes, current psychotic disorder, and current diagnosis of minor or major neurocognitive disorder or suspected neurocognitive disorder with < 24 points on the Mini Mental State Examination number 3, MMSE-NR3.
* ongoing psychotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms using the Montgomery-Asberg Depression Rating Scale, MADRS-S | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  Depressive symptoms measured with the Montgomery-Asberg Depression Rating Self-rating Scale, MADRS-S. MADRS-S is a nine-item questionnaire used to measure severity of depression. The score ranges from 0-54. High scores indicate more depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline in depression diagnosis assessed using the Mini International Neuropsychiatric Interview, MINI | Baseline; Intervention 1 Week 9; 6 months post-intervention.
  MINI is a structured clinical interview used to assess the presence/absence of common psychiatric disorders.
Change from baseline in Physical Activity level | Baseline; Intervention 1 Week 9; 6 months post-intervention.
  Physical Activity levels measured with accelerometer, ActiGraph GT3X. Self rated physical activity levels measured with Frandin/Grimby activity scale, which is a 6 item scale. The score ranges from 0-6. High scores indicate high levels of physical activity.
Change from baseline in anxiety symptoms using the Geriatric Anxiety Scale - 10 item (GAS-10) is a self-rating scale designed to capture anxiety specifically in older adults, with items reflecting affective-, cognitive- and somatic anxiety symptoms. | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  Anxiety symptoms measured with the Geriatric Anxiety Scale -10 version. Self rating symptoms. The score ranges from 0-10. High scores indicate high levels of anxiety.
Change from baseline in health and disability using The WHO Disability Assessment Schedule 12-item, WHODAS | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  WHODAS-12 is a 12-item questionnaire used to assess disability due to health conditions. The total score ranges from 0-48. High scores indicate high levels of disability.
Change from baseline in self rated quality of life using the EuroQol-5 Dimensions-5 Level Scale, EQ-5D-5L | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  The EuroQol-5 Dimensions-5 Level Scale, EQ-5D-5L is a 5-item scale. The scale describes health in five dimensions.
Changes from baseline in Self Efficacy measured with the New General Self-Efficacy Scale, S-GSE. | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  Self efficacy measured with the New General Self-Efficacy Scale, S-GSE. The scale consists of 10 items. Total score ranges from 10-40. High scores indicates high levels of self efficacy.
Changes from baseline in loneliness measured with the UCLA Loneliness Scale version 3, UCLA-LS-3. | Baseline; Intervention 1 Week 9; 3 months post-intervention; 6 months post-intervention.
  Loneliness measured with the UCLA Loneliness Scale version 3, UCLA-LS-3. This is a 20 item scale. Total score ranges from 20-80. High scores indicates low levels of loneliness.
Diagnostic accuracy | Baseline; Week 0
  Area under curve, sensitivity, specificity

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Damberg, MD, Principal Investigator — Uppsala university, Dept. Public Care and Health Sciences
Locations (1):
- Uppsala university, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pellas J, Renner F, Ji JL, Damberg M. Telephone-Based Behavioral Activation with Mental Imagery for Depression in Older Adults in Isolation During the covid-19 Pandemic: Long-term Results from a Pilot Trial. Clin Gerontol. 2023 Jan-Dec;46(5):801-807. doi: 10.1080/07317115.2022.2124899. Epub 2022 Sep 20. PMID 36128612
- [Result] Pellas J, Renner F, Ji JL, Damberg M. Telephone-based behavioral activation with mental imagery for depression: A pilot randomized clinical trial in isolated older adults during the Covid-19 pandemic. Int J Geriatr Psychiatry. 2022 Jan;37(1):10.1002/gps.5646. doi: 10.1002/gps.5646. Epub 2021 Nov 10. PMID 34729823
- [Result] Pellas J, Damberg M. Accuracy in detecting major depressive episodes in older adults using the Swedish versions of the GDS-15 and PHQ-9. Ups J Med Sci. 2021 Oct 20;126. doi: 10.48101/ujms.v126.7848. eCollection 2021. PMID 34754407
- [Derived] Bystrom E, Wennlof B, Johansson I, Lonnberg L, Arkkukangas M, Pellas J, Damberg M. DepActive: study protocol for a randomised controlled multicentre trial of telephone-delivered behavioural activation for the treatment of depression in older adults in primary care. Trials. 2024 Oct 5;25(1):659. doi: 10.1186/s13063-024-08521-y. PMID 39369239